CLINICAL TRIAL: NCT02293252
Title: Gesundheitsökonomische Methodenentwicklung am Beispiel Der Evaluation Einer Technologiebasierten, sektorübergreifenden Intervention Zur Versorgung Chronisch Kranker Patienten
Brief Title: CardioBBEAT - Randomized Controled Trial to Evaluate the Health Economic Impact of Remote Patient Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eckhard Nagel (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Eckhard Nagel, Prof. Dr. Dr. Dr. h.c., University of Bayreuth
Organization: University of Bayreuth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01KX0805
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Heart Failure
Keywords: Home Telemonitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional group (Experimental): Remote patient monitoring system (Motiva)
  Interventions: Device: Remote patient monitoring (Motiva)
- Control group (No Intervention): Best medical treatment according to the guidelines of the European Society of Cardiology (ESC)

INTERVENTIONS:
Device: Remote patient monitoring (Motiva) — interactive bi-directional home telemonitoring system that provides remote monitoring
  Arms: Interventional group

SUMMARY:
The primary endpoint is the incremental cost effectiveness ratio (ICER), defined as the combined clinical endpoint "days alive and not in hospital nor stationary care per days in study" and the change in total cost compared to that of the control group.

DETAILED DESCRIPTION:
Between January 2010 and June 2013, 621 patients with left ventricular ejection fraction (LVEF) ≤ 40% were enrolled and randomly assigned to two study arms comprising usual care and a home telemonitoring group. The 302 patients enrolled in the intervention group are supported by an interactive bi-directional home telemonitoring system (Motiva®) that collects and transfers patient's vital sign data to a dedicated telemedicine data centre. All patients were to remain in the study for one year with an examination at the beginning and both, after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Chronic Heart Failure (CHF) based on European Society of Cardiology (ESC) guidelines
* Symptoms corresponding to New York Heart Association (NYHA) functional class II-IV
* Left Ventricular Ejection Fraction (LVEF) ≤ 40%
* American Heart Association (AHA) classification stage C or D
* Age > 18 years
* Discharged after hospitalisation for worsening Chronic Heart Failure (CHF) within the last twelve months
* Able to understand the German language
* Sufficient eyesight to understand and follow the instructions communicated by the Motiva® platform
* Willing and able to use the required hard- and software and maintain a patient diary
* Residing within geographical reach of one of the ten study sites in order to receive additional treatment if required as well as follow-up consultation
* Willingness to provide informed consent regarding benefits and risks related to the trial, and to sign a participation agreement for the installation of the telemedicine platform Motiva®

Exclusion Criteria:

* Myocardial infarction within the past four weeks
* Heart surgery or any coronary intervention within the past eight weeks
* Cardiogenic shock within the past four weeks
* Intended cardiac surgery within the next six months or priority status on a waiting list for organ transplantation
* Severe chronic and pulmonary illness with an immediate impact on the main outcome measures
* Renal failure requiring dialysis
* Dementia or other severe cognitive impairment
* Psychiatric disorders rendering patients unable to participate in the trial
* Discharged to or living in a geriatric clinic or a nursing home
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2009-03; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
incremental cost effectiveness ratio (ICER) | 1 year
  consisting of the combined clinical endpoint "days alive and not in hospital nor stationary care per days in study" and the change in total cost

SECONDARY OUTCOMES:
Clinical Outcomes - total mortality | 1 year
  total mortality
Clinical Outcome - number of inpatient treatment | 1 year
  number of inpatient treatment
Clinical Outcome - length of stay in hospital or nursing home | 1 year
  length of stay in hospital or nursing home
Clinical Outcome - functional state of health | 1 year
  functional state of health
Clinical Outcome - health related quality of life | 1 year
  health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Nagel, Prof.Dr.mult, Study Chair — Head of Institute for Healthcare Management and Health Science, University of Bayreuth
Locations (1):
- University of Bayreuth, Bayreuth, Bavaria, Germany

REFERENCES:
- [Derived] Voller H, Bindl D, Nagels K, Hofmann R, Vettorazzi E, Wegscheider K, Fleck E, Stork S, Nagel E. The First Year of Noninvasive Remote Telemonitoring in Chronic Heart Failure Is not Cost Saving but Improves Quality of Life: The Randomized Controlled CardioBBEAT Trial. Telemed J E Health. 2022 Mar 21;28(11):1613-22. doi: 10.1089/tmj.2022.0021. Online ahead of print. PMID 35325562
- [Derived] Hofmann R, Voller H, Nagels K, Bindl D, Vettorazzi E, Dittmar R, Wohlgemuth W, Neumann T, Stork S, Bruder O, Wegscheider K, Nagel E, Fleck E; CardioBBEAT Investigators. First outline and baseline data of a randomized, controlled multicenter trial to evaluate the health economic impact of home telemonitoring in chronic heart failure - CardioBBEAT. Trials. 2015 Aug 11;16:343. doi: 10.1186/s13063-015-0886-8. PMID 26259568
- See also: First outline and baseline data of a randomized, controlled multicenter trial to evaluate the health economic impact of home telemonitoring in chronic heart failure - CardioBBEAT — http://www.trialsjournal.com/content/16/1/343